CLINICAL TRIAL: NCT06704269
Title: An Open-label, Multi-center, Phase I/II Study to Assess Safety, Efficacy, and Cellular Kinetics of YTB323 in Participants With Treatment-resistant Generalized Myasthenia Gravis
Brief Title: Study to Assess Safety, Efficacy, and Cellular Kinetics of YTB323 in Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323O12101
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Generalized Myasthenia Gravis
Keywords: myasthenia gravis; generalized myasthenia gravis; YTB323; CAR-T
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YTB323 (Experimental): YTB323 single intravenous (i.v.) infusion
  Interventions: Genetic: YTB323

INTERVENTIONS:
Genetic: YTB323 — CAR-T cell suspension for intravenous infusion

SUMMARY:
This is a phase I/II study to assess safety, efficacy, and cellular kinetics of YTB323 in participants with treatment-resistant generalized myasthenia gravis. YTB323 is a Biological CAR-T cell therapy.

DETAILED DESCRIPTION:
This is an open-label, multi-center, non-confirmatory study intended to assess safety, efficacy, and cellular kinetics of YTB323 treatment in participants with treatment-resistant generalized myasthenia gravis in order to enable a benefit to risk assessment for further development in generalized myasthenia gravis (gMG). The study plans to enroll approximately 15 participants with treatment-resistant gMG. The study utilizes a single dose design across 2 cohorts, consisting of a sentinel cohort of 3 patients followed by an expansion cohort of an additional 12 patients.

All participants dosed with YTB323 will be followed until 15 years after YTB323 administration in the Long-Term Follow-up (LTFU).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed gMG diagnosis supported by the following:

   * Documented report of positive serology testing for either AChR antibodies or MuSK antibodies at screening AND at least one of the following:
   * History of abnormal neuromuscular transmission test demonstrated by repetitive nerve stimulation or single-fiber electromyography
   * History of positive acetylcholinesterase inhibitor test
   * Improvement in MG signs on an oral acetylcholinesterase inhibitor as assessed by the treating physician
2. MGFA Class III-IVa (gMG) at screening
3. Treatment-resistant gMG as defined by: MG-ADL score ≥ 6 (≥50% non-ocular) at screening despite adequate treatment trials with at least two different non-steroidal immunosuppressive drugs given at adequate doses and duration of therapy.
4. If on chronic corticosteroids, must be on a stable dose of corticosteroids for ≥1 month prior to screening and have the ability and willingness to taper to a maximum dose of 10 mg prednisolone daily or equivalent at least one week before leukapheresis
5. If treated with cholinesterase inhibitors, patients must be on a stable dose for at least two weeks prior to screening

Exclusion Criteria:

1. Exclusively ocular myasthenia gravis (MGFA I), mild symptoms (MGFA II), or severe bulbar disease or MG crisis, MGFA Class IVb or V at screening
2. History of bone marrow/hematopoietic stem cell or solid organ transplantation.
3. Clinically significant active, opportunistic, chronic or recurrent infection (including positive for hepatitis B or hepatitis C) confirmed by clinical evidence, imaging, or positive laboratory tests one month prior to leukapheresis
4. Other uncontrolled disease states, such as asthma, or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids, at screening
5. Participants with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug induced immune deficiency), or tested positive for HIV antibody, at screening
6. Prior treatment with anti-CD19 therapy, adoptive T cell therapy or any prior gene therapy product (e.g. CAR-T cell therapy).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2029-10-26 (Estimated); Study Completion 2029-10-26 (Estimated)

PRIMARY OUTCOMES:
Occurrence, severity, and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 2 years
  Incidence of AE's, including Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANs), changes in Vital Signs, Laboratory parameters, ECG, and neurological status qualifying and reported as AEs.

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of YTB323 - CMAX | Pre-dose Day 1 up to 2 years
  Measured by Cmax - The maximum plasma concentration of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - AUC | Pre-dose Day 1 up to 2 years
  Measured by AUC - Area under the curve of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - Tmax | Pre-dose Day 1 up to 2 years
  Measured by Tmax - Time to Reach the Maximum Concentration After Drug Administration of YTB323
Plasma Pharmacokinetics (PK) of YTB323 - Clast | Pre-dose Day 1 up to 2 years
  Clast is defined as the Last observed (quantifiable) plasma concentration (Clast)
Plasma Pharmacokinetics (PK) of YTB323 - Tlast | Pre-dose Day 1 up to 2 years
  Tlast is defined as Time of Last Measurable Concentration
Cellular immunogenicity of YTB323 | Pre-dose lymphodepletion up to 2 years
  Incidence and prevalence of pre-existing and treatment induced humoral immunogenicity of YTB323
Humoral immunogenicity of YTB323 | Pre-dose lymphodepletion up to 2 years
  Incidence and prevalence of pre-existing and treatment induced cellular immunogenicity of YTB323
Neutralizing immunogenicity of YTB323 | Pre-dose lymphodepletion up to 2 years
  Incidence and prevalence of pre-existing and treatment induced neutralizing immunogenicity of YTB323
Change from Baseline of MG-ADL score | Baseline up to 2 years
  The Myasthenia Gravis Activities of Living (MG-ADL) scale is an 8-item patient-reported scale that measures myasthenia gravis symptoms and functional status, to be administered by physician or trained study evaluator. The MG-ADL is an outcome measure assessing MG symptoms and functional activities related to activities of daily living. Each of the items is scored from 0 (normal) to 3 (most severe), providing a total score ranging from 0 to 24, where higher scores indicate greater severity of symptoms. It is composed of items related to patients' assessment of functional disability secondary to ocular (two items), bulbar (three items), respiratory (one item), and gross motor or limb impairment (two items).
Change from Baseline of QMG total score | Baseline up to 2 years
  The Quantitative Myasthenia Gravis (QMG) score is a standardized validated quantitative strength scoring system developed specifically for MG. The QMG is a 13-item direct physician assessment scoring system that quantifies disease severity based on impairments of body functions and structures. Each item is quantitatively assessed and scored from 0 to 3 (where 3 represents the most severe), providing a total QMG score ranging from 0 to 39 where higher scores indicate greater disease activity. The QMG is composed of the following items: ocular (two items), facial (one item), bulbar (two items), gross motor (six items), axial (one item), and respiratory (one item).
Proportion of patients with a ≥3-point reduction of QMG total score sustained for 6 months post Baseline | Baseline up to 2 years
  The QMG score is a standardized validated quantitative strength scoring system developed specifically for MG. The QMG is a 13-item direct physician assessment scoring system that quantifies disease severity based on impairments of body functions and structures. Each item is quantitatively assessed and scored from 0 to 3 (where 3 represents the most severe), providing a total QMG score ranging from 0 to 39, where higher scores indicate greater disease severity. The QMG is composed of the following items: ocular (two items), facial (one item), bulbar (two items), gross motor (six items), axial (one item), and respiratory (one item).
Proportion of patients with a ≥2-point reduction of MG-ADL score sustained for 6 months post Baseline | Baseline up to 2 years
  The Myasthenia Gravis Activities of Living (MG-ADL) scale is an 8-item patient-reported scale that measures myasthenia gravis symptoms and functional status, to be administered by physician or trained study evaluator. The MG-ADL is an outcome measure assessing MG symptoms and functional activities related to activities of daily living. Each of the items is scored from 0 (normal) to 3 (most severe), providing a total score ranging from 0 to 24, where higher scores indicate greater severity of symptoms. It is composed of items related to patients' assessment of functional disability secondary to ocular (two items), bulbar (three items), respiratory (one item), and gross motor or limb impairment (two items).
Proportion of patients with a MGFA-PIS of minimal manifestations (MM) or better and sustained for 6 months post Baseline | Baseline up to 2 years
  The Myasthenia Gravis Foundation of America Post-Intervention Status (MGFA-PIS) is a physician-assessed determination of the overall clinical state of an MG patient at any time after initiation of treatment for MG. MM or better includes Minimal Manifestation (MM): the patient has no symptoms or functional limitations from MG but has some weakness on examination of some muscles; Complete Stable Remission (CSR): the patient has had no symptoms or signs of MG for at least 1 year and has received no therapy for MG during that time. There is no weakness of any muscle on careful examination by someone skilled in the evaluation of neuromuscular disease. Isolated weakness of eyelid closure is accepted; or Pharmacologic Remission (PR): the same criteria as for CSR except that the patient continues to take some form of therapy for MG.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Houston Methodist Hospital, Houston, Texas
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Lille
- Japan (2):
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Kyoto
- United Kingdom (2):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com